CLINICAL TRIAL: NCT06971705
Title: A Study on Precise Cerebral Localization and Network Mechanisms of Repetitive Transcranial Magnetic Stimulation in Treating Chronic Ankle Instability Based on High-resolution Functional Magnetic Resonance Imaging
Brief Title: fMRI Study on Cerebral Localization and Network Mechanisms of rTMS in Chronic Ankle Instability Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Qing Shu, associate chief physician, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025AFD635
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-05

CONDITIONS: Chronic Ankle Instability, CAI; Functional Magnetic Resonance Imaging (fMRI)
Keywords: Chronic ankle instability; functional magnetic resonance imaging; repetitive transcranial magnetic stimulation; ankle stability training
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding After the intervention allocation, the participants and data analysts will be blinded. This is a single - blinded, randomized, parallel - controlled study focusing on rTMS. In the real rTMS group, a 10 - minute magnetic stimulation will be applied to the target brain area. The sham stimulation can imitate the sensation of real stimulation without causing any physiological effects. Before the final code - breaking, data analysts won't know the group to which the data they are analyzing belongs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham rTMS plus ankle stability training (Placebo Comparator)
  Interventions: Behavioral: ankle stability training; Device: Sham repetitive transcranial magnetic stimulation, SrTMS
- rTMS plus ankle stability training (Experimental)
  Interventions: Device: repetitive transcranial magnetic stimulation, rTMS; Behavioral: ankle stability training

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation, rTMS — Participants underwent rTMS intervention prior to daily ankle stability training. The interventional targets were the key cortical brain regions identified in preliminary studies, with stimulation applied to the contralateral cortical areas corresponding to the affected ankle joint. Parameters included a figure-of-8 coil, 10 Hz frequency, 2-second stimulation duration, 8-second inter-train intervals, 60 repetitions, totaling 1,200 pulses per session, with each session lasting 10 minutes. Ankle stability training commenced within 10 minutes post-rTMS, following the same duration and intensity as the Ankle Stability Training Group + Sham rTMS Group. The treatment was conducted three times per week for a total of 4 weeks.
  Arms: rTMS plus ankle stability training
Behavioral: ankle stability training — The ankle stability training protocol comprised three modalities: neuromuscular training, balance training, and proprioceptive training. Specific exercises included single-leg stance, balance pad training, heel raises, resistive ankle inversion/eversion exercises, MOBO board balance exercises, alphabet tracing (toe-writing), lateral walking, heel walking, toe walking, and jump and landing control drills. The training progressed from stable to unstable surfaces, starting at low intensity and gradually increasing in difficulty and intensity. The training was conducted three times per week for a total of 4 weeks.
Device: Sham repetitive transcranial magnetic stimulation, SrTMS — Before each session of ankle stability training, participants received sham rTMS intervention. The sham stimulation mimicked the sensory experience of real rTMS but did not produce any physiological effects.
  Arms: Sham rTMS plus ankle stability training

SUMMARY:
Chronic ankle instability (CAI) is a common sports injury that often leads to recurrent injuries and functional deficits. While conventional rehabilitation can restore ankle stability, the underlying neurophysiological mechanisms remain poorly understood, and the long-term efficacy of current treatments is limited. This study aims to investigate the therapeutic efficacy of repetitive transcranial magnetic stimulation (rTMS) in combination with conventional ankle stability training for CAI and to evaluate its impact on ankle-stabilizing muscle activation and cerebral cortex excitability.

The study design is a single-center, randomized, single-blind, parallel-controlled trial. Participants with CAI will be randomly assigned to either an ankle stability training plus real rTMS group or an ankle stability training plus sham rTMS group. The primary outcome measure is the Cumberland Ankle Instability Tool (CAIT) score, which assesses the severity of ankle instability. Secondary outcomes include the Karlsson-Peterson Ankle Function Score (KPAFS), American Orthopedic Foot and Ankle Society Score (AOFAS), surface electromyography (sEMG) data, and task-based functional magnetic resonance imaging (fMRI) data. These secondary outcomes will provide a comprehensive evaluation of ankle function, muscle activation patterns, and neural activity changes.

The intervention will consist of a 4-week program, with participants receiving rTMS sessions three times per week. Each rTMS session will target key brain regions. The ankle stability training will include exercises designed to improve strength, balance, and proprioception. The sham rTMS group will receive identical ankle stability training but with a placebo rTMS protocol to ensure blinding.

Data will be collected at baseline, 2 weeks, and 4 weeks. The primary outcome, CAIT score, will be used to assess the overall improvement in ankle stability. The KPAFS and AOFAS scores will provide additional measures of ankle function and pain. sEMG data will be collected during specific functional tasks to evaluate the activation patterns of the tibialis anterior, peroneus longus, and other relevant muscles. Task-based fMRI will be used to assess changes in brain activity in motor and sensory areas before and after the intervention.

Statistical analyses will be performed using SPSS 22.0. Data will be presented as mean ± standard deviation. Between-group differences will be compared using independent samples t-tests, and overall differences across time points will be assessed via two-way repeated-measures ANOVA or mixed-effects models. Post-hoc analyses will be conducted to identify specific time points and conditions where significant differences occur.

The study timeline spans from March 2025 to December 2026, including participant recruitment, intervention implementation, data collection, and analysis, as well as manuscript drafting. This research aims to provide new insights into the neurophysiological mechanisms of CAI and to offer a novel, evidence-based approach to the rehabilitation of CAI, potentially improving long-term outcomes and reducing the risk of recurrent injuries.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years.
2. History of at least one significant ankle sprain within the past 12 months, accompanied by inflammatory response (including pain resulting in at least one day of restricted physical activity).
3. The most recent ankle sprain must have occurred more than 3 months prior to enrollment.
4. Self-reported symptoms of ankle instability, defined by one or more of the following: At least two episodes of "giving way" in the affected ankle within the past 6 months; Recurrent sprains (≥2 documented sprains in the same ankle); Subjective perception of instability confirmed by any one of the following validated instruments: Ankle Instability Instrument (AII): ≥5 affirmative responses; Cumberland Ankle Instability Tool (CAIT): Score <24; Identification of Functional Ankle Instability (IdFAI): Score >11.
5. Foot and Ankle Ability Measure (FAAM): Activities of Daily Living (ADL) subscale <90%; FAAM Sports subscale <80%; Foot and Ankle Outcome Score (FAOS): Scores <75% in ≥3 subcategories.

Exclusion Criteria:

1. Chronic ankle instability caused by bilateral ankle sprains;
2. History of lower extremity musculoskeletal or neurological surgery;
3. History of lower extremity fractures;
4. Acute musculoskeletal injuries in other lower extremity joints within 3 months that compromised joint integrity and function, resulting in ≥1 day of interrupted daily or sports activities;
5. Concomitant severe systemic diseases (cardiac, pulmonary, hepatic, renal, etc.);
6. Severe psychiatric disorders or cognitive impairments;
7. Presence of metal implants or inability to tolerate MRI examinations.
8. Patient refusal to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Cumberland Ankle Instability Tool score, CAIT | Before treatment, 2 week after treatment and 4 weeks after treatment
  A self-reported questionnaire designed to assess functional ankle instability. It consists of 9 items with a total score ranging from 0 to 30, where higher scores indicate better ankle stability.

SECONDARY OUTCOMES:
Karlsson-Peterson Ankle Function Score, KPAFS | Before treatment, 2 week after treatment and 4 weeks after treatment
  The KPAFS is a scoring system used to evaluate ankle dysfunction. It includes 10 items: pain, daily activities, walking ability, need for support, squatting ability, ankle range of motion, limb positioning, limb length, limb circumference, and limb appearance. Each item is scored based on the patient's condition, with a total possible score of 100. Higher scores indicate better ankle function.
American Orthopedic Foot and Ankle Society score, AOFAS | Before treatment, 2 week after treatment and 4 weeks after treatment
  The AOFAS is a widely used assessment tool for evaluating functional outcomes in foot and ankle disorders. It includes domains such as pain, function, gait, range of motion, stability, and foot alignment. The total score ranges from 0 to 100, with higher scores reflecting better foot and ankle function.
Surface electromyography | Before treatment and 4 weeks after treatment
  The surface electromyography of the tibialis anterior, gastrocnemius, and peroneus longus muscles was tested while the subjects were standing on one leg and undergoing the star excursion balance test (SEBT). The following indicators were collected:
  1. Time-domain analysis indicators: Root Mean Square (RMS), Integrated Electromyography (iEMG), and Averaged Electromyography (AEM).
  2. Frequency-domain analysis indicators: Mean Power Frequency (MPF) and Median Frequency (MF).
fMRI | Before treatment and 4 weeks after treatment
  Task - related fMRI data were collected by using the affected lower limb isometric contraction combined with "single - leg standing" motor imagery.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan hospital of Wuhan University, Wuhan, Hubei, China

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT06971705/Prot_SAP_000.pdf